CLINICAL TRIAL: NCT07128212
Title: Atorvastatin Mitigates WMH-Related Cognitive Impairment by Reducing VCAM-1: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Atorvastatin Mitigates WMH-Related Cognitive Impairment by Reducing VCAM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Municipal Hospital of Anhui Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SuzhouAnhuiWMH
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ischemic White Matter Lesions (WMIL); Cerebral Small Vessel Disease; Vascular Cell Adhesion Molecule-1; VCAM-1
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WMH - Intervention (Experimental): Participants with WMH receiving oral atorvastatin 10 mg once daily at 18:00 (6 p.m.) for 24 months. Standard assessments will be performed at baseline and follow-up.
  Interventions: Drug: Atorvastatin 10 mg daily
- WMH - Placebo (Placebo Comparator): Participants with WMH receiving a placebo tablet matching atorvastatin, administered orally once daily at 18:00 (6 p.m.) for the same duration as the intervention arm. The same assessments will be performed.
  Interventions: Drug: Placebo matching atorvastatin
- Health Control (No Intervention): Health control participants with no study intervention; baseline and follow-up assessments only over the same schedule as patient groups.

INTERVENTIONS:
Drug: Atorvastatin 10 mg daily — Oral atorvastatin 10 mg administered once daily at 18:00 (6 p.m.) for 24 months. Dose form: tablet. Route: oral. Indicated for participants with WMH. Adherence monitored by pill count and diary. No dose titration planned.
  Other Names: Atorvastatin calcium; ATV
  Arms: WMH - Intervention
Drug: Placebo matching atorvastatin — Placebo tablet matching atorvastatin in appearance and packaging, containing inactive excipients only; taken orally once daily at 18:00 for 24 months.
  Arms: WMH - Placebo

SUMMARY:
This prospective study will enroll patients younger than 60 years with ischemic white matter lesions (WMIL) and age-matched healthy controls. We will measure circulating endothelial-related biomarkers, including endothelial progenitor cells (EPCs), intercellular adhesion molecule-1 (ICAM-1), vascular cell adhesion molecule-1 (VCAM-1), asymmetric dimethylarginine (ADMA), and homocysteine (Hcy). We will also assess transcription levels of ICAM-1, VCAM-1, and ADMA. All participants will be followed and managed for 2 years, with repeated assessments of endothelial biomarkers and their transcriptional levels, as well as clinical and imaging evaluations. The aims are to characterize changes in endothelial biomarkers in WMIL, to determine how these changes relate to clinical features and imaging progression, and to evaluate whether statins protect endothelial function-by modifying these biomarkers-and thereby help treat WMIL and slow its progression.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-60 years.
* Provides written informed consent.
* WMIL group: consecutive outpatients/inpatients from the Neurology Department of Suzhou Municipal Hospital, with WMIL confirmed by brain MRI. Diagnostic features: symmetric, diffusely distributed, ill-defined lesions in periventricular and subcortical white matter; iso- or hypointense on T1WI; hyperintense on T2WI and FLAIR.
* Control group: healthy individuals aged 45-60 years with brain MRI showing no intracranial lesions.

Exclusion Criteria:

* Acute intracerebral hemorrhage or acute infarction on brain MRI or CT.
* Central nervous system diseases that severely affect cognition, such as Alzheimer's disease or frontotemporal dementia.
* White matter lesions due to other causes (e.g., toxic, genetic, immune, infectious, neoplastic, radiation-related).
* Severe hepatic, renal, or cardiac insufficiency.
* Recent major surgery or severe trauma.
* History of psychiatric disorders that would preclude completion of study scales.
* Unable to provide written informed consent.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
VACM1 levels at 0.5, 1.0, 1.5, and 2.0 years | 0.5, 1, 1.5, and 2.0 years after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hospital of Anhui Medical University, Suzhou, Anhui, China